CLINICAL TRIAL: NCT02333240
Title: Self-management of Postnatal Anti-hypertensive Treatment: a Trial Development Pilot Study
Acronym: SNAP-HT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10959
Record Dates: First submitted 2014-12-15; First posted 2015-01-07 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-05

CONDITIONS: Pre-Eclampsia; Hypertension, Pregnancy-Induced
Keywords: Pregnancy; Postnatal Care; Blood Pressure Monitoring, Home; Self Care; Pregnancy Complications, Cardiovascular; Qualitative Research; Antihypertensive Agents
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced; Pregnancy Complications, Cardiovascular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual care (No Intervention): Women randomised to usual care will have their blood pressure monitored by their community midwife, and will have their anti-hypertensive medication adjusted by their general practitioner. There will be no intervention in this group.
  All women will be followed up at ten days, four and six weeks, then three and six months postpartum and have their blood pressure measured by one of the study team.
- Self-management (Experimental): Self-management of postnatal anti-hypertensive treatment. Women will be provided with, and taught to use, a validated home blood pressure monitor, and perform daily BP readings. When treatment is discontinued we will ask them to continue daily BP measurements for 1 week. Provided these are <140/90 mmHg they will be asked to check their BP weekly for the remainder of the trial period. The self-monitoring BP data will be collated centrally through the use of a smart phone app or SMS based system. This service will respond to participants regarding the level of their BP and what action is required. Women in the self-management group will have an individualised medication adjustment schedule developed by the research team in conjunction with the participant's obstetric team.
  Interventions: Other: Self-management of postnatal anti-hypertensive treatment

INTERVENTIONS:
Other: Self-management of postnatal anti-hypertensive treatment — Daily use of a validated home blood pressure monitor in conjunction with an individualised medication adjustment schedule to adjust anti-hypertensive medications in line with blood pressure readings.
  Arms: Self-management

SUMMARY:
New-onset raised blood pressure (BP) affects about one in ten pregnancies. For some women, raised BP is an indication of pre-eclampsia: newly arising high blood pressure in pregnancy combined with protein leaking into the urine. After birth, women's BP remains elevated for a period of time, but in most cases returns to normal over 2-12 weeks. During this period medication needs to be adjusted to achieve the correct control. Research suggests that better BP control during this period is associated with improved long-term health outcomes. The investigators would like to find out whether home BP monitoring, and self-adjustment of medications according to an individualised protocol, could improve BP control and patient satisfaction.

This pilot study has been set up to inform the planning of a large-scale multi-centre randomised controlled trial by testing the feasibility of the protocol. The investigators want to increase our experience of applying this management approach in this subset of patients; to select the most appropriate primary outcome measure and to estimate the effect size of this intervention; to assess recruitment potential; and to evaluate feasibility of coordinating this trial across several centres. The primary objective of the large-scale trial will be to determine whether the self-management approach can improve BP control in women with medicated hypertensive disorders of pregnancy in the postnatal period.

Women recruited to the study will be randomly assigned to one of two groups: self-management or usual care. Participants allocated to 'usual care' will have their BP monitored and medication adjusted by their general practitioner (GP) and midwife as normal. Participants allocated to the 'self-management' group will use a home BP monitor daily following discharge from hospital after birth. They will be provided with an individualised schedule for gradually decreasing their medication(s) in line with their BP readings. Women will be followed up for 6 months.

DETAILED DESCRIPTION:
Hypertensive disorders of pregnancy (HDP) affect 3-15% of pregnancies. Gestational hypertension is new-onset blood pressure (BP) > 140/90mmHg after 20 weeks gestation. Pre-eclampsia is gestational hypertension with proteinuria (> 300mg / 24 hours). HDP are the second commonest direct cause of maternal death in the UK and USA, and the leading cause of maternal death in Latin America and the Caribbean.

HDP persist postpartum, and complications can occur during this time. Most women with HDP will be treatment-free by 3 months postpartum. This rapidly changing BP, with shifting medication requirement, poses a challenge in terms of how best to manage this down-titration. Both NICE guidelines and a Cochrane review highlight that few clinical studies have addressed the management of BP postpartum. In practice clinical care is to continue antepartum anti-hypertensive medication and monitor BP in the community with a focus on prevention of over-treatment.

Approximately 30% of eclamptic seizures occur postpartum: studies suggest that half occur more than 48 hours after birth. A case series of patients who sustained a stroke in association with HDP, showed that more than half occurred postpartum.

Severity of hypertension in later life may be predicted by BP during the first 6 weeks postpartum. Several retrospective cohort studies and a meta-analysis have suggested that HDP are associated with an increased risk of future cardiovascular disease (CVD) in the mother. The 2011 American Heart Association guidelines for the prevention of CVD in women cite a history of HDP as a major risk factor for CVD, and advocate enquiring about pregnancy complications during the evaluation of CVD risk.

Home BP readings have been shown to be more strongly related to indices of target organ damage and have better prognostic value in essential hypertension than office BP measurement. Voluntary home BP monitoring by patients with essential hypertension is becoming increasingly common. The European and American Societies of Hypertension now recommend home BP measurement in the routine diagnosis and monitoring of essential hypertension.

Self-monitoring and self-titration of anti-hypertensive medications in essential hypertension has been shown to be both feasible and more effective than usual care. Women with HDP would seem to be an ideal cohort in whom to apply these experiences: the disease has, in general, a limited time course meaning that intensive monitoring is more reasonable and more likely to be adhered to. Pregnant women are in a younger age group than the majority of those with essential hypertension, and may be more comfortable with the use of technology to assist in disease monitoring. Women might also be more empowered in the setting of a recent pregnancy to take greater responsibility for their health.

Evidence exists to support the accuracy of home BP recordings in hypertensive pregnant women. Studies to date in antenatal women suggest a low non-concordance rate and low rate of inaccurate recordings. Studies have also suggested: better correlation between home BP recordings and indication of the need for anti-hypertensive medication; reduced number of hospital admissions in women with mild HDP who undertook home BP monitoring.

If self-management in the postpartum period proves to be feasible, acceptable and successful, it could lead to a reduction in the length of inpatient stay, readmissions and the number of postpartum visits, with cost-saving implications. Furthermore as the importance of BP control in the immediate postpartum period has already been demonstrated to affect women's CVD risk up to 15 years after delivery, any strategy, which successfully increases women's adherence to an effective treatment regimen, has the potential to influence their healthcare needs well into the future.

The proposed trial aims to apply the research experience regarding self-management in essential hypertension to postpartum women with HDP where both high and low BPs can lead to adverse outcomes, and where detection of on-going hypertension is essential. This study is a pilot study: it has been set up in order to inform the planning of a large-scale multi-centre randomised controlled trial by testing the feasibility of methods and procedures for later use on a large scale. We want to increase our experience of applying this management approach in this subset of patients; to select the most appropriate primary outcome measure and to estimate the effect size of this intervention; to assess recruitment potential; and to evaluate the feasibility of coordinating this trial across several centres. The primary objective of the large-scale trial will be to determine whether the self-management approach can improve BP control in women with medicated HDP in the postnatal period.

The study is a non-blinded randomised controlled trial. To assist with recruitment numbers, and assess the feasibility of running a multi-centre trial, we are planning to run this study in several hospitals. Women who have developed HDP requiring medication will be approached during the antenatal period: they will complete an informed consent form and undertake a screening appointment. Following birth, whilst they remain in hospital, consent will be confirmed and a baseline appointment will take place. At this visit women will be randomised to one of two treatment arms: usual care, or self-management.

All women will be followed up at 10 days, 4 and 6 weeks, then 3 and 6 months postpartum and have their BP measured by one of the study team. All participants will be asked to complete the EQ-5D-5L Health Questionnaire to assess their quality of life at visits 1, 5 and 7.

At visits 2, 6 and 7 women will be weighed using a standardised set of scales in order to evaluate whether the extent and speed of return to booking weight correlates with resolution of gestational hypertension.

To follow on from the work that suggests that those with above-average BP at six weeks postpartum have an approximately 30% increase in aortic stiffness, we are planning to conduct a sub-study to analyse markers of vascular risk in women from both groups. As it may be assumed that the baseline characteristics of the two groups are then similar, if we demonstrate a treatment effect from the intervention, then it will allow us to analyse the relationship between BP control in the postnatal period and markers of vascular risk to help determine if it is the severity of pathology or effectiveness of control that determines long term outcome. Women will consent to an optional extended visit at baseline and 3 months where measures of arterial stiffness and microvascular changes will be taken (cardio-ankle vascular index, radial arterial tonometry and capillaroscopy). We will take a blood sample to measure circulating biomarkers relevant to cardiovascular health and pre-eclampsia. We aim to recruit a minimum of 15 women from each group.

We plan to run a second embedded sub-study to examine participants' health experiences. We aim to recruit a minimum of 50% of participants in each group. We will conduct structured interviews with participants in both arms, who consent to participate in the qualitative sub-study, to assess their experience of either usual care or self-management of BP in the postnatal period, and to identify and explore factors related to the successful (or unsuccessful) implementation of the intervention. This study will provide data regarding the views of patients as to the acceptability of self-monitoring in the routine management of gestational hypertension and pre-eclampsia after birth once they have been discharged from hospital. Baseline data (5 questions) will be collected at visit 1. The structured interviews will be done at visits 4 and 7, and will take 10-15 minutes on each occasion. There will be 5 questions for both groups, and an additional 5 questions for the intervention group. Structured responses will be entered on to a pre-coded scoring sheet. Free text responses will be audio-recorded.

Safety reporting will be from baseline to the 26 week follow up visit. Adverse events may be recorded by the participant using the trial telephone number, email, or via the text message service or smart phone app. Participants will be directly asked about adverse events at each study visit. All serious adverse events, whether 'expected' or 'unexpected', need to be reported. All serious adverse event (SAE) information will be recorded on the Primary Care Clinical Trials Unit (PC-CTU) SAE report form by the site or the Chief Investigator (CI) and faxed to the PC-CTU dedicated fax line. SAEs will be reported to the PC-CTU as soon as possible, preferably within 24 hours. The PC-CTU will perform an initial check of the report, request any additional information from the reporting clinician and ensure that the CI or safety delegator reviews and evaluates the report for expectedness and relatedness. All SAE reports will also be reviewed routinely by the Independent Safety Review Committee. All SAEs will be followed up until resolution or the end of the study period.

A SAE occurring to a participant should be reported to the REC and Sponsor where in the opinion of the Chief Investigator the event was 'related' (resulted from administration of any of the research procedures) and 'unexpected' in relation to those procedures. Reports of related and unexpected SAEs should be submitted within 15 working days of the CI becoming aware of the event.

A formal sample size calculation is not required for this pilot study. The analysis will be carried out on the basis of intention-to-treat. The analyses for this pilot study will be primarily descriptive and will not include any hypothesis testing or presentation of P-values for group comparisons. Continuous variables will be reported as means with standard deviations (or medians with Interquartile ranges if skewed). Categorical variables will be reported as counts and percentages. Differences between groups will be calculated and described with 95% confidence intervals only and will not include significance tests with P-values.

The delivery of the intervention will involve patient home visits. To facilitate these visits the study team will require access to patient identifiable data. The consent from will clearly list the data to be collected and for what purpose. The identifiable data will be held securely at the PC-CTU, separately from other trial data, with access to this data restricted to appropriate members of the study team identified on the delegation log. Identifiable data will be anonymised as soon as no longer required.

All study data required for analysis will be recorded on paper Case Report Forms (CRFs) and returned to the study team for data entry. CRFs will be held securely in locked filing cabinets, located within office space with restricted entry. All data points will be transferred from paper CRFs to a secure database management system (CDMS) hosted by the PC-CTU. Within the CDMS patients will be identified solely by a unique study identification number. No patient identifiable data will be held within the CDMS. At the conclusion of the trial, following database lock and final analysis all documents will be appropriately archived for at least five years.

The CI will ensure the study is conducted in accordance with the current approved protocol, PC-CTU SOPs and all applicable local and national guidelines and regulations. The PC-CTU has conducted a risk assessment prior to study commencement, which will inform the level and nature of monitoring required for this study. Direct access will be granted to authorised representatives from the Sponsor or host institution for monitoring and/or audit of the study to ensure compliance with regulations.

A Trial Management Group will be established to support the CI in overseeing the progress and conduct of the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Female, aged 18 years or above.
* Women with gestational hypertension (new-onset BP > 140/90mmHg) or pre-eclampsia (new onset BP > 140/90mmHg and significant proteinuria > 300mg/24hr), prior to their discharge from hospital post-delivery.
* Require antihypertensive medication during pregnancy, which needs to continue in the postpartum period.

Exclusion Criteria:

* Hypertension prior to pregnancy.
* Poor English language skills.
* More than three anti-hypertensive agents at discharge from hospital postpartum.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2015-04; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Feasibility: recruitment rate | 13 months from trial start date (end of the recruitment period)
  Number of participants randomised / number of consenting participants Number of participants randomised / number of potential participants approached
Feasibility: retention rate | Up to 19 months from trial start date
  Number of participants completing trial follow up / number of participants randomised
Feasibility: attrition rate | Up to 19 months from trial start date
  Number of participants lost to follow-up or withdrawn / number of participants randomised
Feasibility: compliance rate | Up to 19 months from trial start date
  Number of study visits attended / total number of intended study visits

SECONDARY OUTCOMES:
Mean systolic blood pressure at follow up visits | 6 months from baseline visit
  Mean of systolic blood pressure at day 10, 4 weeks, 6 weeks, 12 weeks and 26 weeks postpartum Number of blood pressure readings in target range 'Time to event': number of urgent visits, and timing of these, to GP or hospital requiring medication increase due to BP > 150/100, or medication decrease due to BP < 100 systolic
Mean diastolic blood pressure at follow up visits | 6 months from baseline visit
  Mean of diastolic blood pressure at day 10, 4 weeks, 6 weeks, 12 weeks and 26 weeks postpartum Number of blood pressure readings in target range 'Time to event': number of urgent visits, and timing of these, to GP or hospital requiring medication increase due to BP > 150/100, or medication decrease due to BP < 100 systolic
Change in participant self-assessed quality of life from screening visit to 6 week follow up visit | 6 weeks from baseline visit
  Change in EQ-5D-5L health questionnaire results from screening visit to 6 week follow up Structured interviews (participants) EQ-5D-5L health questionnaire results Structured interviews (participants)
Change in participant self-assessed quality of life from screening visit to 6 month follow up visit | 6 months from baseline visit
  Change in EQ-5D-5L health questionnaire results from screening visit to 6 month follow up Structured interviews (participants) EQ-5D-5L health questionnaire results Structured interviews (participants)
Change in cardio-ankle vascular index from baseline to 3 months | 3 months from baseline visit
  Cardio-ankle vascular index
Change in pulse wave velocity from baseline to 3 months | 3 months from baseline visit
  Radial arterial tonometry
Change in capillary density from baseline to 3 months | 3 months from baseline visit
  Microvascular changes: capilloroscopy
Change in laboratory values from baseline to 3 months | 3 months from baseline visit
  Haemoglobin, platelets, creatinine, alanine transferase, uric acid, lipid profile, insulin, glucose and novel markers of pre-eclampsia
Safety (reporting adverse events and side effects) | 6 months from baseline visit
  Reporting of serious adverse events Reporting of side effects

OTHER OUTCOMES:
To explore percentage time spent in range as a marker for blood pressure control in this setting. (percentage time spent in target BP range) | 6 months from baseline visit
  Assess percentage time spent in target BP range in both groups, and use the home monitoring data from the intervention arm to explore the validity of this measure and the relationship between the trial blood pressure readings taken at two time points
Setting BP thresholds for future trials (Difference between home and clinic BP recordings) | 6 months from baseline visit
  Difference between home and clinic BP recordings

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra E Cairns, BMBCh MA, Principal Investigator — Nuffield Department of Primary Care Health Sciences, University of Oxford
Locations (5):
- United Kingdom (5):
  - Royal Berkshire NHS Foundation Trust, Reading, Berkshire
  - Northampton General Hospital NHS Trust, Northampton, Northamptonshire
  - Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire
  - Stoke Mandeville Hospital, Aylesbury
  - Horton General Hospital, Banbury

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ananth CV, Keyes KM, Wapner RJ. Pre-eclampsia rates in the United States, 1980-2010: age-period-cohort analysis. BMJ. 2013 Nov 7;347:f6564. doi: 10.1136/bmj.f6564. PMID 24201165
- [Background] Cantwell R, Clutton-Brock T, Cooper G, Dawson A, Drife J, Garrod D, Harper A, Hulbert D, Lucas S, McClure J, Millward-Sadler H, Neilson J, Nelson-Piercy C, Norman J, O'Herlihy C, Oates M, Shakespeare J, de Swiet M, Williamson C, Beale V, Knight M, Lennox C, Miller A, Parmar D, Rogers J, Springett A. Saving Mothers' Lives: Reviewing maternal deaths to make motherhood safer: 2006-2008. The Eighth Report of the Confidential Enquiries into Maternal Deaths in the United Kingdom. BJOG. 2011 Mar;118(Suppl 1):1-203. doi: 10.1111/j.1471-0528.2010.02847.x. PMID 21356004
- [Background] Khan KS, Wojdyla D, Say L, Gulmezoglu AM, Van Look PF. WHO analysis of causes of maternal death: a systematic review. Lancet. 2006 Apr 1;367(9516):1066-1074. doi: 10.1016/S0140-6736(06)68397-9. PMID 16581405
- [Background] Walters BN, Walters T. Hypertension in the puerperium. Lancet. 1987 Aug 8;2(8554):330. doi: 10.1016/s0140-6736(87)90912-3. No abstract available. PMID 2886783
- [Background] Podymow T, August P. Postpartum course of gestational hypertension and preeclampsia. Hypertens Pregnancy. 2010;29(3):294-300. doi: 10.3109/10641950902777747. PMID 20670153
- [Background] Chames MC, Livingston JC, Ivester TS, Barton JR, Sibai BM. Late postpartum eclampsia: a preventable disease? Am J Obstet Gynecol. 2002 Jun;186(6):1174-7. doi: 10.1067/mob.2002.123824. PMID 12066093
- [Background] Martin JN Jr, Thigpen BD, Moore RC, Rose CH, Cushman J, May W. Stroke and severe preeclampsia and eclampsia: a paradigm shift focusing on systolic blood pressure. Obstet Gynecol. 2005 Feb;105(2):246-54. doi: 10.1097/01.AOG.0000151116.84113.56. PMID 15684147
- [Background] Lazdam M, de la Horra A, Diesch J, Kenworthy Y, Davis E, Lewandowski AJ, Szmigielski C, Shore A, Mackillop L, Kharbanda R, Alp N, Redman C, Kelly B, Leeson P. Unique blood pressure characteristics in mother and offspring after early onset preeclampsia. Hypertension. 2012 Nov;60(5):1338-45. doi: 10.1161/HYPERTENSIONAHA.112.198366. Epub 2012 Oct 8. PMID 23045462
- [Background] Magee L, von Dadelszen P. Prevention and treatment of postpartum hypertension. Cochrane Database Syst Rev. 2013 Apr 30;2013(4):CD004351. doi: 10.1002/14651858.CD004351.pub3. PMID 23633317
- [Background] Mosca L, Benjamin EJ, Berra K, Bezanson JL, Dolor RJ, Lloyd-Jones DM, Newby LK, Pina IL, Roger VL, Shaw LJ, Zhao D, Beckie TM, Bushnell C, D'Armiento J, Kris-Etherton PM, Fang J, Ganiats TG, Gomes AS, Gracia CR, Haan CK, Jackson EA, Judelson DR, Kelepouris E, Lavie CJ, Moore A, Nussmeier NA, Ofili E, Oparil S, Ouyang P, Pinn VW, Sherif K, Smith SC Jr, Sopko G, Chandra-Strobos N, Urbina EM, Vaccarino V, Wenger NK. Effectiveness-based guidelines for the prevention of cardiovascular disease in women--2011 update: a guideline from the american heart association. Circulation. 2011 Mar 22;123(11):1243-62. doi: 10.1161/CIR.0b013e31820faaf8. Epub 2011 Feb 14. No abstract available. PMID 21325087
- [Background] Ray JG, Vermeulen MJ, Schull MJ, Redelmeier DA. Cardiovascular health after maternal placental syndromes (CHAMPS): population-based retrospective cohort study. Lancet. 2005 Nov 19;366(9499):1797-803. doi: 10.1016/S0140-6736(05)67726-4. PMID 16298217
- [Background] Wilson BJ, Watson MS, Prescott GJ, Sunderland S, Campbell DM, Hannaford P, Smith WC. Hypertensive diseases of pregnancy and risk of hypertension and stroke in later life: results from cohort study. BMJ. 2003 Apr 19;326(7394):845. doi: 10.1136/bmj.326.7394.845. PMID 12702615
- [Background] Lykke JA, Langhoff-Roos J, Sibai BM, Funai EF, Triche EW, Paidas MJ. Hypertensive pregnancy disorders and subsequent cardiovascular morbidity and type 2 diabetes mellitus in the mother. Hypertension. 2009 Jun;53(6):944-51. doi: 10.1161/HYPERTENSIONAHA.109.130765. Epub 2009 May 11. PMID 19433776
- [Background] McDonald SD, Malinowski A, Zhou Q, Yusuf S, Devereaux PJ. Cardiovascular sequelae of preeclampsia/eclampsia: a systematic review and meta-analyses. Am Heart J. 2008 Nov;156(5):918-30. doi: 10.1016/j.ahj.2008.06.042. Epub 2008 Oct 2. PMID 19061708
- [Background] Paradisi G, Biaggi A, Savone R, Ianniello F, Tomei C, Caforio L, Caruso A. Cardiovascular risk factors in healthy women with previous gestational hypertension. J Clin Endocrinol Metab. 2006 Apr;91(4):1233-8. doi: 10.1210/jc.2005-1337. Epub 2006 Jan 24. PMID 16434462
- [Background] Stergiou GS, Bliziotis IA. Home blood pressure monitoring in the diagnosis and treatment of hypertension: a systematic review. Am J Hypertens. 2011 Feb;24(2):123-34. doi: 10.1038/ajh.2010.194. Epub 2010 Sep 9. PMID 20940712
- [Background] Bobrie G, Chatellier G, Genes N, Clerson P, Vaur L, Vaisse B, Menard J, Mallion JM. Cardiovascular prognosis of "masked hypertension" detected by blood pressure self-measurement in elderly treated hypertensive patients. JAMA. 2004 Mar 17;291(11):1342-9. doi: 10.1001/jama.291.11.1342. PMID 15026401
- [Background] Baral-Grant S, Haque MS, Nouwen A, Greenfield SM, McManus RJ. Self-Monitoring of Blood Pressure in Hypertension: A UK Primary Care Survey. Int J Hypertens. 2012;2012:582068. doi: 10.1155/2012/582068. Epub 2011 Oct 16. PMID 22013510
- [Background] Little P, Barnett J, Barnsley L, Marjoram J, Fitzgerald-Barron A, Mant D. Comparison of acceptability of and preferences for different methods of measuring blood pressure in primary care. BMJ. 2002 Aug 3;325(7358):258-9. doi: 10.1136/bmj.325.7358.258. No abstract available. PMID 12153924
- [Background] Parati G, Stergiou GS, Asmar R, Bilo G, de Leeuw P, Imai Y, Kario K, Lurbe E, Manolis A, Mengden T, O'Brien E, Ohkubo T, Padfield P, Palatini P, Pickering T, Redon J, Revera M, Ruilope LM, Shennan A, Staessen JA, Tisler A, Waeber B, Zanchetti A, Mancia G; ESH Working Group on Blood Pressure Monitoring. European Society of Hypertension guidelines for blood pressure monitoring at home: a summary report of the Second International Consensus Conference on Home Blood Pressure Monitoring. J Hypertens. 2008 Aug;26(8):1505-26. doi: 10.1097/HJH.0b013e328308da66. PMID 18622223
- [Background] Pickering TG, Miller NH, Ogedegbe G, Krakoff LR, Artinian NT, Goff D; American Heart Association; American Society of Hypertension; Preventive Cardiovascular Nurses Association. Call to action on use and reimbursement for home blood pressure monitoring: executive summary: a joint scientific statement from the American Heart Association, American Society Of Hypertension, and Preventive Cardiovascular Nurses Association. Hypertension. 2008 Jul;52(1):1-9. doi: 10.1161/HYPERTENSIONAHA.107.189011. Epub 2008 May 22. PMID 18497371
- [Background] McManus RJ, Mant J, Bray EP, Holder R, Jones MI, Greenfield S, Kaambwa B, Banting M, Bryan S, Little P, Williams B, Hobbs FD. Telemonitoring and self-management in the control of hypertension (TASMINH2): a randomised controlled trial. Lancet. 2010 Jul 17;376(9736):163-72. doi: 10.1016/S0140-6736(10)60964-6. Epub 2010 Jul 8. PMID 20619448
- [Background] McManus RJ, Mant J, Haque MS, Bray EP, Bryan S, Greenfield SM, Jones MI, Jowett S, Little P, Penaloza C, Schwartz C, Shackleford H, Shovelton C, Varghese J, Williams B, Hobbs FD, Gooding T, Morrey I, Fisher C, Buckley D. Effect of self-monitoring and medication self-titration on systolic blood pressure in hypertensive patients at high risk of cardiovascular disease: the TASMIN-SR randomized clinical trial. JAMA. 2014 Aug 27;312(8):799-808. doi: 10.1001/jama.2014.10057. PMID 25157723
- [Background] Waugh J, Habiba MA, Bosio P, Boyce T, Shennan A, Halligan AW. Patient initiated home blood pressure recordings are accurate in hypertensive pregnant women. Hypertens Pregnancy. 2003;22(1):93-7. doi: 10.1081/PRG-120017007. PMID 12648446
- [Background] Rayburn WF, Zuspan FP, Piehl EJ. Self-monitoring of blood pressure during pregnancy. Am J Obstet Gynecol. 1984 Jan 15;148(2):159-62. doi: 10.1016/s0002-9378(84)80168-4. PMID 6691392
- [Background] Barton JR, Stanziano GJ, Sibai BM. Monitored outpatient management of mild gestational hypertension remote from term. Am J Obstet Gynecol. 1994 Mar;170(3):765-9. doi: 10.1016/s0002-9378(94)70279-9. PMID 8141198
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Background] Lancaster GA, Dodd S, Williamson PR. Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract. 2004 May;10(2):307-12. doi: 10.1111/j..2002.384.doc.x. PMID 15189396
- [Background] Rosendaal FR, Cannegieter SC, van der Meer FJ, Briet E. A method to determine the optimal intensity of oral anticoagulant therapy. Thromb Haemost. 1993 Mar 1;69(3):236-9. PMID 8470047
- [Derived] Kitt JA, Fox RL, Cairns AE, Mollison J, Burchert HH, Kenworthy Y, McCourt A, Suriano K, Lewandowski AJ, Mackillop L, Tucker KL, McManus RJ, Leeson P. Short-Term Postpartum Blood Pressure Self-Management and Long-Term Blood Pressure Control: A Randomized Controlled Trial. Hypertension. 2021 Aug;78(2):469-479. doi: 10.1161/HYPERTENSIONAHA.120.17101. Epub 2021 Jun 28. PMID 34176288
- [Derived] Cairns AE, Tucker KL, Crawford C, McManus RJ, Powell J. Implementing self-management: a mixed methods study of women's experiences of a postpartum hypertension intervention (SNAP-HT). Trials. 2020 Jun 9;21(1):508. doi: 10.1186/s13063-020-04394-z. PMID 32517785
- [Derived] Cairns AE, Tucker KL, Leeson P, Mackillop LH, Santos M, Velardo C, Salvi D, Mort S, Mollison J, Tarassenko L, McManus RJ; SNAP-HT Investigators. Self-Management of Postnatal Hypertension: The SNAP-HT Trial. Hypertension. 2018 Aug;72(2):425-432. doi: 10.1161/HYPERTENSIONAHA.118.10911. Epub 2018 Jul 2. PMID 29967037
- See also: NICE Clinical Guideline 107 (Hypertension in pregnancy) — http://www.nice.org.uk/guidance/CG107